CLINICAL TRIAL: NCT00784147
Title: A Phase 2b, Randomized, Double-Blinded, 48-Week, Multicenter, Dose-Response Study of Ibalizumab Plus an Optimized Background Regimen in Treatment-Experienced Patients Infected With HIV-1(Amended to 24-Weeks)
Brief Title: Dose-Response Study of Ibalizumab (Monoclonal Antibody) Plus Optimized Background Regimen in Patients With HIV-1
Acronym: TMB-202
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: TaiMed Biologics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TMB-202 Amendment 2
Record Dates: First submitted 2008-10-30; First posted 2008-11-03 (Estimated); Results first posted 2014-04-17 (Estimated); Last update posted 2014-05-05 (Estimated); Status verified 2014-04

CONDITIONS: HIV
Keywords: HIV; CD4; experienced; resistant; resistance; monoclonal; antibody; infusion; ibalizumab; TNX355; TNX-355; TMB355; TMB-355
MeSH Terms: interventions — ibalizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ibalizumab 800 mg (Active Comparator): every 2 weeks, combined with an Optimized Background Regimen
  Interventions: Drug: Ibalizumab
- Ibalizumab 2000 mg (Active Comparator): every 4 weeks, combined with an Optimized Background Regimen
  Interventions: Drug: Ibalizumab

INTERVENTIONS:
Drug: Ibalizumab — Ibalizumab 800 mg IV every 2 weeks
  Other Names: TNX-355; Hu5A8
  Arms: Ibalizumab 800 mg
Drug: Ibalizumab — Ibalizumab 2000 mg IV every 4 weeks
  Other Names: TNX-355; Hu5A8
  Arms: Ibalizumab 2000 mg

SUMMARY:
The investigational product, ibalizumab, is a humanized IgG4 monoclonal antibody administered via intravenous infusion at 800 mg every 2 weeks or at 2000 mg every 4 weeks. In addition to study drug, all patients will receive an optimized background regimen (OBR), which is a standard-of-care regimen selected by the investigator prior to randomization that is comprised of 2-4 antiretroviral agents. These agents must have been approved by the local regulatory agency or be available through expanded-access programs for treatment of human immunodeficiency virus (HIV).

DETAILED DESCRIPTION:
The primary objectives of this study are to:

* Evaluate the dose-response relationship of antiviral activity of the ibalizumab dose regimens at Week 24 in order to determine the optimal dose and regimen. The primary evaluation of effectiveness will be based on the proportion of patients achieving undetectable viral loads at Week 24.
* Evaluate the safety and tolerability of two dose regimens of ibalizumab for dose selection

The secondary objectives of this study are to:

* Evaluate changes from Baseline in viral load, CD4+ cell counts, and time to loss of virologic response (TLOVR)
* Characterize HIV-1 sensitivity/susceptibility changes associated with ibalizumab administration in combination with OBR
* Determine the presence and significance of anti-ibalizumab antibodies, if any (immunogenicity of ibalizumab)
* Assess CD4 receptor density and occupancy
* Determine the impact of ibalizumab on quality of life as assessed by patient-reported outcomes on questionnaires
* Evaluate the pharmacokinetic profile of two dose regimens of ibalizumab at steady state

ELIGIBILITY:
Inclusion Criteria:

1. Are capable of understanding and have voluntarily signed the informed consent document
2. Have documented HIV-1 infection by official, signed, written history (eg, laboratory report), otherwise an HIV-antibody test will be performed
3. Have no acquired immunodeficiency syndrome (AIDS)-defining events in the 3 months before screening, other than cutaneous Kaposi's sarcoma or wasting syndrome due to HIV
4. Are able and willing to comply with all protocol requirements and procedures
5. Are 18 years of age or older
6. Have a life expectancy that is >6 months.
7. Have a viral load >1,000 copies/mL and documented decreased susceptibility to at least one NRTI, one NNRTI, and one PI, as measured by resistance testing
8. Are receiving a stable highly active antiretroviral regimen for at least 8 weeks before screening and are willing to continue that regimen until the baseline visit, OR (in the past 8 weeks) have failed and are off therapy and are willing to stay off therapy until the baseline visit
9. Have viral sensitivity/susceptibility to at least one agent (OSS criteria) as determined by the screening resistance tests and be willing and able to be treated with at least one agent to which the patient's viral isolate is sensitive/susceptible according to the screening resistance tests as a component of OBR
10. If sexually active, are willing to use an effective method of contraception during the study and for 30 days after the last administration of the study drug

Exclusion Criteria:

1. Any active AIDS-defining illness per Category C conditions according to the Center for Disease Control (CDC) Classification System for HIV Infection, with the following exceptions: cutaneous Kaposi's sarcoma and wasting syndrome due to HIV
2. Any significant diseases (other than HIV-1 infection) or clinically significant findings, including psychiatric and behavioral problems, determined from screening, medical history and/or physical examination that, in the investigator's opinion, would preclude the patient from participating in this study
3. Any significant acute illness within 1 week before the initial administration of study drug
4. Any active infection secondary to HIV requiring acute therapy; however, patients that require maintenance therapy (ie, secondary prophylaxis for opportunistic infections) will be eligible for the study
5. Any immunomodulating therapy (including interferon), systemic steroids, or systemic chemotherapy within 12 weeks before randomization
6. Any investigational therapy within 30 days before randomization, except for HIV-agents available in expanded-access programs
7. Any prior exposure to ibalizumab (formerly TNX-355 and Hu5A8)
8. Any vaccination within 21 days before randomization
9. Any female patient who either is pregnant, intends to become pregnant, or is currently breast-feeding
10. Any current alcohol or illicit drug use that, in the investigator's opinion, will interfere with the patient's ability to comply with the study schedule and protocol evaluations
11. Any previous clinically significant allergy or hypersensitivity to any excipient in the ibalizumab formulation
12. Any radiation therapy during the 28 days before first administration of investigational medication
13. Any grade 3 or 4 toxicity according to the Division of AIDS grading scale, except for the following asymptomatic grade 3 events: triglyceride elevation & total cholesterol elevation

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 113 (Actual)
Dates: Start 2008-08; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stanley T. Lewis, MD, Study Director — TaiMed Biologics Inc.
Locations (30):
- United States (28):
  - AIDS Health Care Foundation - Research, Beverly Hills, California
  - Living Hope Clinical Foundation, Long Beach, California
  - Kaiser Permanente Medical Center, Los Angeles, California
  - Quest Clinical Research, San Francisco, California
  - Kaiser Permanente Medical Center Research Unit, San Francisco, California
  - Kaiser Permanente of Colorado, Denver, Colorado
  - National Jewish Medical & Research Center, Denver, Colorado
  - Whitman-Walker Clinic, Washington D.C., District of Columbia
  - South Florida Clinical Research, Atlantis, Florida
  - University of Miami, Miller School of Medicine, Miami, Florida
  - Orlando Immunology Center, Orlando, Florida
  - Associates in Infectious Diseases, Port Saint Lucie, Florida
  - Treasure Coast Infectious Disease Consultants, Vero Beach, Florida
  - Triple O Medical Services, Inc., West Palm Beach, Florida
  - Northstar Medical Center, Chicago, Illinois
  - Indiana University School of Medicine - Wishard Memorial Hospital, Indianapolis, Indiana
  - St. Michael's Medical Center, Newark, New Jersey
  - AIDS Community Research Initiative of America, New York, New York
  - The Brody School of Medicine at ECU, Greenville, North Carolina
  - The Research & Educational Group, Portland, Oregon
  - Central Texas Clinical Research, Austin, Texas
  - North Texas Infectious Disease Consultants, Dallas, Texas
  - Valley AIDS Council, Harlingen, Texas
  - Therapeutic Concepts, Houston, Texas
  - University of Texas Health Science Center, Houston, Texas
  - Nationsmed Clinical Research, Houston, Texas
  - Dr. Gordon E. Crofoot, MD, PA, Houston, Texas
  - Research Access Network, Houston, Texas
- Puerto Rico (2):
  - Clinical Research Puerto Rico, San Juan
  - HOPE Clinical Research, San Juan

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Over the period from late 2008 through early 2010, a total of 113 patients were enrolled into the study from 35 study sites in the United States and Taiwan. The study sites were private medical practices, not-for-profit community clinics and university hospital clinics delivering HIV primary care.
Groups:
- Ibalizumab 800 mg: every 2 weeks, combined with an Optimized Background Regimen
  Ibalizumab : Ibalizumab 800 mg IV every 2 weeks
- Ibalizumab 2000 mg: every 4 weeks, combined with an Optimized Background Regimen
  Ibalizumab : Ibalizumab 2000 mg IV every 4 weeks
Period: Overall Study
Arm/Group | Ibalizumab 800 mg | Ibalizumab 2000 mg
Started | 59 | 54
Completed | 51 | 45
Not Completed | 8 | 9
Not completed — Lost to Follow-up | 2 | 4
Not completed — Withdrawal by Subject | 1 | 3
Not completed — Physician Decision | 2 | 1
Not completed — Protocol Violation | 1 | 1
Not completed — Death | 2 | 0

BASELINE CHARACTERISTICS:
Population: Baseline measures were assessed using the Intent-to-Treat (ITT) population, defined as all randomized patients regardless of whether a dose of study medication was received.
Groups:
- Total: Total of all reporting groups
Arm/Group | Ibalizumab 800 mg | Ibalizumab 2000 mg | Total
Number analyzed (Participants) | 59 | 54 | 113
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 58 | 54 | 112
  >=65 years | 1 | 0 | 1
Age, Continuous [Mean (Full Range); unit: years] | 48.3 [29.6 to 69.5] | 47.9 [32.6 to 62.3] | 48.1 [29.6 to 69.5]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 4 | 12
  Male | 51 | 50 | 101
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 3 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 12 | 15 | 27
  White | 42 | 28 | 70
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 4 | 8 | 12
HIV-1 RNA (viral load) [Mean (Full Range); unit: copies/mL] | 114,675.3 [58.0 to 1,087,333.3] | 136,452.8 [1,893.3 to 1,573,333.3] | 125,082.2 [58.0 to 1,573,333.3]
CD4+ T-cell count [Mean (Standard Deviation); unit: cells/mL] | 106.4 (91.3) | 112.4 (118.5) | 109.3 (104.7)
Number of active agents in OBR [Mean (Standard Deviation); unit: Pharmaceutical Agents] | 1.9 (0.8) | 1.8 (0.7) | 1.8 (0.7)
Time from initial documented HIV infection [Mean (Standard Deviation); unit: years] — Time elapsed from initial documentation of HIV infection - when known - to the first administration of study drug. This information was available and recorded for slightly less than half of the study participants (N = 52).
  years | 17.0 (4.4) | 16.9 (6.2) | 17.0 (5.4)

OUTCOME MEASURES:

1. Primary Outcome: The Proportion of Patients Achieving Undetectable Viral Loads at Week 24.
Description: For the primary efficacy analysis, "undetectable" was defined as having HIV-1 RNA below the limit of assay detection at <50 copies/mL. The primary efficacy endpoint was analyzed using Fisher exact test. The primary analysis was performed using the ITT population and both the missing data equals treatment failure (MEF) and last observation carried forward (LOCF) methods. The more conservative MEF results are recorded here.
Time Frame: 24 weeks
Measure: Number; unit: percentage of participants
Arm/Group | Ibalizumab 800 mg | Ibalizumab 2000 mg
Number analyzed (Participants) | 59 | 54
percentage of participants | 44 | 28

2. Other Pre Specified Outcome: Proportion of Patients With Viral Load <200 Copies/mL at Week 24
Description: This measure was assessed in the same manner as the primary efficacy analysis for the proportion of patients achieving HIV-1 RNA levels below 200 copies/mL at Week 24 of the study.
Time Frame: Week 24
Measure: Number; unit: percentage of patients
Arm/Group | Ibalizumab 800 mg | Ibalizumab 2000 mg
Number analyzed (Participants) | 59 | 54
percentage of patients | 53 | 43

3. Other Pre Specified Outcome: Proportion of Patients With Viral Load <400 Copies/mL at Week 24
Description: This efficacy measure was assessed in the same manner as the primary efficacy analysis to determine the proportion of the total population achieving HIV-1 RNA levels <400 copies at Week 24 of the study.
Time Frame: Week 24
Measure: Number; unit: percentage of patients
Arm/Group | Ibalizumab 800 mg | Ibalizumab 2000 mg
Number analyzed (Participants) | 59 | 54
percentage of patients | 58 | 46

4. Other Pre Specified Outcome: Proportion of Patients With a 1.0 log10 or Greater Reduction in Viral Load at Week 24
Description: This efficacy assessment was performed in the same manner as the primary efficacy analysis for the proportion of the total population achieving at least a 1.0 log10 reduction from Baseline in HIV-1 RNA.
Time Frame: Week 24
Measure: Number; unit: percentage of patients
Arm/Group | Ibalizumab 800 mg | Ibalizumab 2000 mg
Number analyzed (Participants) | 59 | 54
percentage of patients | 63 | 59

5. Other Pre Specified Outcome: Proportion of Patients With a 0.5 log10 or Greater Reduction in Viral Load at Week 24
Description: This efficacy assessment was performed in the same manner as the primary efficacy analysis for the proportion of the total population achieving at least a 0.5 log10 reduction from the Baseline measurement in HIV-1 RNA at Week 24 of the study.
Time Frame: Week 24
Measure: Number; unit: percentage of patients
Arm/Group | Ibalizumab 800 mg | Ibalizumab 2000 mg
Number analyzed (Participants) | 59 | 54
percentage of patients | 68 | 59

6. Secondary Outcome: Mean Change From Baseline in Viral Load (log10) at Week 24/EOS
Description: The mean change in HIV-1 RNA (log10) from the Baseline measurement was analyzed at Week 24/End of Study using a generalized linear model at each scheduled study visit.
Time Frame: Week 24 / End of Study
Measure: Mean (Standard Deviation); unit: log10 copies/mL
Arm/Group | Ibalizumab 800 mg | Ibalizumab 2000 mg
Number analyzed (Participants) | 59 | 54
log10 copies/mL | -1.6 (1.3) | -1.5 (1.4)

7. Secondary Outcome: Mean Change From Baseline in CD4+ T-Cell Count at Week 24/EOS
Description: The mean change in CD4+ T-cell count from the Baseline measurement at Week 24/End of Study was summarized at each scheduled time point by treatment group.
Time Frame: Week 24 / End of Study
Measure: Mean (Standard Deviation); unit: cell/mL
Arm/Group | Ibalizumab 800 mg | Ibalizumab 2000 mg
Number analyzed (Participants) | 59 | 54
cell/mL | 36.5 (63.0) | 39.8 (80.1)

ADVERSE EVENTS:
Time Frame: Through Week 24 of the Study
Arm/Group | Ibalizumab 800 mg | Ibalizumab 2000 mg
Serious Adverse Events (participants affected / at risk) | 7/59 | 3/54
Other Adverse Events (participants affected / at risk) | 46/59 | 44/54
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ibalizumab 800 mg (N=59) | Ibalizumab 2000 mg (N=54)
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — Moderate Severity Unrelated to Study Drug Administration
Acute Renal Failure (Renal and urinary disorders) | 1 (1) | 0 (0) — Severe. Unrelated to Study Drug Administration
Gastroenteritis (Gastrointestinal disorders) | 1 (1) | 0 (0) — Severe. Unrelated to Study Drug Administration.
Road Traffic Accident (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) — Life-threatening. Unrelated to Study Drug Administration.
Paraesthesias (Nervous system disorders) | 1 (1) | 0 (0) — Moderate. Unrelated to Study Drug Administration.
Cerebral Toxoplasmosis (Infections and infestations) | 0 (0) | 1 (1) — Moderate. Unrelated to Study Drug Administration.
CMV Viremia (Infections and infestations) | 0 (0) | 2 (3) — One instance of moderate severity, two severe occurrences. Unrelated to Study Drug Administration.
Acute Respiratory Distress Syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — Fatal. Unrelated to Study Drug Administration
End-stage AIDS (Immune system disorders) | 1 (1) | 0 (0) — Fatal. Unrelated to Study Drug Administration.
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ibalizumab 800 mg (N=59) | Ibalizumab 2000 mg (N=54)
Rash (Skin and subcutaneous tissue disorders) | 5 (5) | 9 (9)
Diarrhea (Gastrointestinal disorders) | 3 (3) | 6 (6)
Nausea (Gastrointestinal disorders) | 2 (2) | 7 (7)
Upper Respiratory Tract Infection (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 3 (3)
Headache (General disorders) | 2 (2) | 4 (4)
Fatigue (General disorders) | 3 (3) | 3 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 0 (0)
Oral Candidiasis (Infections and infestations) | 2 (2) | 4 (4)
Nasopharyngitis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3)
Dizziness (General disorders) | 4 (4) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 3 (3)
Sinusitis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Folliculitis (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (3)
Low Back Pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2)
Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)
Chills (General disorders) | 1 (1) | 2 (2)
Conjunctivitis (Eye disorders) | 1 (1) | 2 (2)
Injection Site Reaction (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Rhinitis Allergic (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)

LIMITATIONS AND CAVEATS:
ACTG Adherence Questionnaire data were incomplete due to insufficient data collection methods. No clinically meaningful information was gained upon review of these results.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less